CLINICAL TRIAL: NCT05825157
Title: Prospective Evaluation of Combination Therapy for Upper Extremity Lymphedema
Brief Title: Evaluation of Combination Therapy for Upper Extremity Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Dung Nguyen, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67367
Record Dates: First submitted 2022-11-29; First posted 2023-04-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lymphedema Arm

STUDY DESIGN:
Intervention Model Description: VLNT or VLNT with BioBridge placement
Who Masked: Participant
Masking Description: patients will be blinded and be randomized via a blocked randomization design. Approximately 60 patients will be randomized in a 4:1 ratio to the intervention arm (VLNT + BioBridge): control arm (VLNT alone). Randomization will be done within blocks (of size 5) so that the balance between treatments is preserved throughout the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- VLNT (Active Comparator): Standard of care vascularized lymph node transfer
  Interventions: Device: BioBridge
- VLNT with Biobridge (Experimental): Standard of care vascularized lymph node transfer plus BioBridge placement
  Interventions: Device: BioBridge

INTERVENTIONS:
Device: BioBridge — Fibralign BioBridge is a thread-like, multi-lumen scaffold consisting of highly aligned collagen fibrils, optimized to encourage the endothelial cell attachment,alignment and migration that are prerequisites to new vessel formation. BioBridge is a device made from highly purified, medical-grade porcine collagen.

SUMMARY:
Investigate whether the addition of the Biobridge scaffold to the standard surgery for vascularized lymph node transfer will improve the outcome of surgical treatment in lymphedema of the upper extremity. Will Biobridge improve upon the low success rate of the currently practiced surgery by facilitating the lymphatic connections to the transplanted node that are crucial to its viability and function.

DETAILED DESCRIPTION:
Secondary lymphedema is the most common cause of lymphedema in the western world. Vascularized lymph node transfer (VLNT) is currently practiced with increasing frequency in the human disease population. This study will determined the efficacy of the Biobridge when used with VLNT in the human subjects with lymphedema; efficacy in large animal models has already been demonstrated. Patients with lymphedema who had BioBridge placed for soft tissue reinforcement after scar release has been observed to have improved lymph drainage and improvement of their limb volume.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 75 years (inclusive)
* Life expectancy > 2 years
* Upper limb lymphedema
* The participant must be eligible for surgical intervention
* Swelling of 1 limb that is not completely reversed by elevation or compression
* Stage I-II lymphedema at screening, based on the International Society of Lymphology (ISL) staging system
* Participants with a history of cancer must have no evidence of disease (NED), have completed breast cancer therapy 3 years prior to enrollment; use of endocrine therapy is allowed.
* Completion of a full course of complete decongestive therapy (CDT), according to ISL guidelines at least 12 weeks prior to screening, including use of compression garments for at least 12 weeks without change in regimen
* Willingness to comply with recommended regimen of self care, with consistent use of compression garments from screening through the entire study duration (through the safety follow up visit), excluding the first 3 weeks postoperatively where patients are required to not wear compression. Self bandaging, use of nighttime compression garments, and intermittent pneumatic compression devices are allowed, but the procedures and regimens are expected to remain consistent from screening though the entire study duration.
* Consistent use of an appropriately sized compression garment for daytime use.
* Limb volume (LV) in the affected limb and unaffected limb must be at least 10% of each other.
* Evidence of abnormal bioimpedance ratio, if feasible, based upon unilateral disease: L Dex > 10 units.
* Willingness and ability to comply with all study procedures, including measurement of limb volume, skin biopsy, and preoperative and postoperative imaging studies.
* Willingness and ability to understand, and to sign a written informed consent form document

Exclusion Criteria:

* Edema arising from increased capillary filtration will be excluded (venous incompetence).
* Inability to safely undergo general anesthesia and/or perioperative care related to vascularized lymph node transfer
* Concurrent participation in a clinical trial of any other investigational drug or therapy, regardless of indication, within 1 month before screening or 5 times the drug's half life, whichever is longer
* Recent initiation (≤ 12 weeks) of CDPT for lymphedema
* Other medical condition that could lead to acute limb edema, such as (but not limited to) acute venous thrombosis or heart failure
* Other medical condition that could result in symptoms overlapping those of lymphedema in the affected limb (e.g., pain, swelling, decreased range of motion)
* History of clotting disorder (hypercoagulable state)
* Chronic (persistent) infection in the affected limb
* Infection of the lymphedema limb within 1 month prior to screening
* Currently receiving chemotherapy or radiation therapy
* Body Mass Index (BMI) >35
* Known sensitivity to porcine products
* Anaphylaxis to iodine
* Pregnancy or nursing
* Substance abuse (such as alcohol or drug abuse) within 6 months prior to screening
* Any reason (in addition to those listed above) that, in the opinion of the investigator, precludes full participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Improve the outcome of surgical treatment of upper extremity lymphedema | 12 months
  To measure the post-surgical percent change in excess limb volume measured at 12 months following surgery using BioBridge scaffold as an adjunct to vascularized lymph node transfer for treatment of upper extremity lymphedema
Improve the outcome of surgical treatment of upper extremity lymphedema | 12 months
  Primary endpoint is % change in (excess) limb volume, from baseline to Month 12, in the intervention group relative to control group. Dispersion (variance) will be assessed as the standard deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No